CLINICAL TRIAL: NCT06614413
Title: Randomized Controlled Clinical Trial: Dietetic-nutritional Intervention Based on the Mediterranean Diet During Pregnancy and the First Two Years, First Thousand Days, for the Improvement of Neurological Development
Brief Title: Intervention Based on the Mediterranean Diet During Pregnancy and the First Two Years for the Improvement of Neurological Development
Acronym: CONMED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Esperanza Escribano, Pediatrician; Neonatologist, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HULP/6812; PI24/0035 (Other Grant/Funding Number: Proyectos Acción Estratégica en Salud)
Record Dates: First submitted 2024-09-19; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Diet, Mediterranean; Pregnancy Related; Child Development; Infant Behaviour

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mother-child binomial with nutritional intervention (Active Comparator): Interventions will be based on dietary-nutritional advice, derived from scientific evidence: nutrition based on the Mediterranean diet (MD) and usual treatment
  Interventions: Other: Neurodevelopment and behaviour assesment 2 years old
- Mother-child binomial as a control group (with follow-up without intervention). (Placebo Comparator): Mother-child binomial as a control group, with follow-up without intervention.
  Interventions: Other: Neurodevelopment and behaviour assesment 2 years old

INTERVENTIONS:
Other: Neurodevelopment and behaviour assesment 2 years old — Mothers: Monthly visits guided or not by nutritionist (intervention vs control group) will consist in food questionnaires and 3-day food diary collection during pregnancy. Every three months during lactation. Children: From one year of age onwards, the KIDMED questionnaire will be administered quarterly Neurodevelopment and behavior assessment 18-24 months of age

SUMMARY:
The main objective is to evaluate the effect of the Mediterranean diet during pregnancy and the first two years of the child&#39;s life on the child&#39;s neurodevelopment and behavior (externalizing and internalizing disorders) measured at one and a half and two years. Secondary objectives are to evaluate the effect of the Mediterranean diet on: body composition at two years of age in infants (densitometry) and of the mother at 3 months postpartum, the incidence of allergic disease in infants, the fetal and infant ́s growth and metabolic risk in the mother during pregnancy and in the boy/girl at two years (fasting glucose: insulin, HOMA), LDL and HDL cholesterol, and micronutrient status (iron, calcium, phosphorus, magnesium, sodium, potassium, chloride, selenium, zinc and LCPUFAs).

Randomized controlled clinical trial with a 1:1 ratio, parallel and open label. Group 1: Mother-child binomial with nutritional intervention; Group 2: Mother-child binomial as a control group (with follow-up without intervention).

Assuming a loss of 25% (10% at follow-up, 15% failure of nutritional intervention) we would need a sample size of 267 patients per group. 1. Evaluation of neurodevelopment using the Bayleys scale version -III, at 2 years of age. 2.

Behavioral assessment CBCL at 1.5 and two years and BRIEF-P at two years.

DETAILED DESCRIPTION:
It will be registered in ClinicalTrials.gov. Randomization will be carried out in blocks of 50 patients (the last of 34 for having a total of 534 patients).

using the "sample" function of the statistical program R version 4.0.2 (R Core Team, 2020).

Study subjects:

All adult pregnant women who attend the routine first trimester visit from 4 weeks + 0 days of gestation up to 14 weeks + 6 days of gestation will be candidates to participate in the study.

The study will be carried out at the La Paz University Hospital, and in associated health centers.

Estimation of sample size:

1. Using the cognitive development score of the Bayleys III test at 2 years: A sample size of 200 patients per group reaches a power of 80% to reject the null hypothesis of equality of means when the difference in population means is μ1 - μ2 = 123.6 - 118.6 = 5.0 with a standard deviation of 17.8 for both groups (JAMA Netw Open. 2023) and with a significance level (alpha) of 0.05 using a two-sample t test of equal variances.
2. Using the socioemotional score of the Bayleys III test: A sample size of 200 patients per group (for the diet and control group) reaches a power of 80% to reject the null hypothesis of equality of means when the difference in population means is μ1 - μ2 = 108.6 - 103.4 = 5.2 with a standard deviation of 18.5 for both groups (JAMA Netw Open. 2023) and with a significance level (alpha) of 0.05 using a two-way t test samples of equal variances.

Assuming a loss of 25% (10% at follow-up, 15% failure of nutritional intervention) we would need a sample size of 267 patients per group.

The sample size estimate is smaller using CBCL with two repeated measures for the outcome variables.The number of women recruited with a statistical power of 0.8 and an alpha value of 0.5 should be 82 infants per group. Assuming losses of 25%, a total of 107 per group.

In order to objectively evaluate adherence to the MEDITERRANEAN diet (MD), the following will be used:

* Quantification of total phenolic compounds (CFT) in urine samples: The total phenolic compounds will be determined in urine samples. For the determination of total phenolic compounds in urine, a procedure will be followed. Spectrophotometric method using the Folin-Ciocalteu reagent, described and validated by Medina-Remón et al. We will perform a solid phase pre-extraction using OASIS 30 mg MAX 96-well plates to remove interferences with the Folin-Ciocalteu reagent. For the determination of CFT, the gallic acid will be used as a reference. Creatinine will be determined using a method previously described (Jaffé M. et al.) and adapted for plates of 96 wells by Medina-Remón et al. A calibration curve will be prepared for creatinine. CFTs will be normalized by creatinine and will be expressed as mg equivalents of gallic acid/g of creatinine.
* Magnetic resonance, analysis of metabolic fingerprints and biomarkers of specific food intake and food groups, precise measurement, developed and validated at Imperial College London (doi:10.1016/S2213-8587(16)30419-3, 10.1038/s43016-020-0093-y).

Study variables:

1. Bayleys scale version III deriving the following four scales (raw and typical scalar derived scores): (a) cognitive, (b) language (receptive and expressive), (c) motor (fine and gross), and (d) socioemotional.
2. Evaluation of behavior, externalizing problems in the child (attention deficit, aggressiveness) and internalizing disorders (anxiety, depression) through validated parent surveys. For this they will be used:

   * Child Behavior Checklist (CBCL), parents will answer this questionnaire.
   * BRIEF-P (Behavior Rating Inventory for Executive Function-Preschool), which is an instrument designed to evaluate executive function (EF) of infants, as an endophenotypic indicator of externalizing problems, after two years. From this test the following three indices will be extracted:
   * Inhibitory self-control index,
   * Flexibility Index
   * Emergent metacognition index. A psychologist, accredited for Bayleys III, will carry out the neurodevelopmental evaluation and the questionnaires will be evaluated, as well as the Bayleys test blind to the child's group.
3. Evaluation of secondary objectives, influence of MD:

3.1. Micronutrient status in the child. They are related to the nutritional status of infants and may have a significant impact on the development and health of the nervous system. Blood determinations of:

* Omega-3 fatty acids, especially docosahexaenoic acid (DHA).
* Iron.
* Vitamin D and retinol transport protein.
* Calcium, phosphorus, magnesium, selenium, and zinc. 3.2. Additionally, blood samples will be used for proteomics and evaluation of epigenetic changes (the latter also in the father).

3.3. Body composition: the measurement of body composition will be carried out using DEXA (X-ray absorptiometry dual energy). This very low dose X-ray technique determines body composition considering 3 components: lean tissue, fat and bone. The values obtained allow the calculation of fat mass indices (IMG) and lean (IMM) as indicators of nutritional status (Mazess RB et. al. 1990). The densitometry will acquire software in the GE IDXA Lunar Densitometer: enCORE v17, installed in the Nuclear Medicine Service from the La Paz University Hospital. 3.4. Oxidative damage to proteins, lipids and DNA in urine. 3.5. Composition of breast milk, given that it has been observed that dietary intake can modify the composition of breast milk (BM), milk samples will be collected from mothers during the lactation period (at 3 months postpartum).

3.6. Microbiota. To know the relationship that MD adherence has with changes in the microbiota of mothers and infants, analysis of feces, milk and vaginal exudate will be performed in the mother and feces in the child for measurement of microbiota and analysis of short-chain fatty acids in feces.

Data collection:

In the mother:

1. Sociodemographic data of the mother (age, highest level of education achieved, employment situation and status socioeconomic (monthly net salary of the family unit), country of birth, street of residence to estimate minimum average income and environmental pollution.
2. Obstetric history: gestational diabetes, weight gain, first, second and third trimester, diseases associated with pregnancy.
3. Maternal prenatal history: body mass index, pregestational diabetes.
4. During pregnancy: Fasting glucose/insulin, HOMA; blood pressure, anemia in mother, maternal medication.
5. Data on mothers' physical activity practice in the third trimester of pregnancy through Pregnancy Physical Activity Questionnaire (PPAQ)
6. Type of delivery.
7. Postpartum: Abdominal waist measurement and body composition (% fat mass and lean mass) at 3 months delivery.
8. Type of breastfeeding.
9. Toxic habits: smoker before, during pregnancy and breastfeeding. Ingestion of alcohol or other toxic substances before, during pregnancy and breastfeeding.

In the infant-toddler:

1. Sex, weight, length and head circumference at birth, 3, 9, 18 and 24 months and dietary diary at 6, 12, 18 and 24 months of age.
2. Incidence of allergic disease: Diagnoses of atopic dermatitis, asthma, recurrent bronchospasm and presence of food allergies at 6, 12, 18 and 24 months.
3. Quality of life at two years old as reported by parents using the TAPQOL questionnaire.
4. Micronutrient values .
5. Body composition at two years measured by densitometry.
6. Use of screens evaluated using the SCREENQ, a questionnaire completed by parents.
7. Health assessment (including events and medications).
8. Number of siblings and position (1st, 2nd...).
9. Exposure to green areas. All questionnaires will be used in their Spanish version.

Statistical analysis The statistical study will be carried out at the end of the study by intention to treat. Good adhesion is defined by protocol such as improvement in three points in the 17-food questionnaire in mothers. As the main variable is in toddlers, we will consider good adherence to the DM in these according to the questionnaire score KIDMED at 24 months: ≥8 good adherence; 4-7 intermediate adhesion; ≤3 low adhesion. As possible confounding variables, the effect of breastfeeding, defined as exclusive (≥ 6 months of age), mixed (< 6 months of breastfeeding with the use of formula) or artificial breastfeeding; the sex of the child and the socioeconomic level of the families defined as the net monthly income of the family unit (<€1,300; €1300 - €1900; €1900 - €2550; €2550 - €3550; €3550 - €4500; >€4500).

The description of the qualitative data will be done in the form of absolute frequencies and percentages and the data quantitative using mean and standard deviation or median and interquartile range, depending on the distribution of this data.

The normality of the continuous variables will be studied using the Kolmogorov Smirnov test.

For the comparison between the diet groups and the qualitative variables, the Pearson Chi-Square test will be used.

For the target variables, measured after two years, that show differences according to the diet groups, generalized linear models to adjust the effect of diet for the variables considered to be confounding described previously. All statistical tests will be considered bilateral and as significant values, those p lower 0.05.

ELIGIBILITY:
1. Inclusion Criteria:

   a. Fluency in the Spanish language, singleton pregnancy
2. Exclusion Criteria:

   1. Children conceived with assisted reproduction techniques
   2. Fetal anomalies and congenital infections
   3. Neonatal anomalies diagnosed after birth
   4. Intellectual development disorder, due to clinical judgment, inability to attend visits
   5. Participation in another controlled trial
   6. Vegetarian diet

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnants
Enrollment: 534 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Neurodevelopmental assessment an behavior at 2 years old | Assessment at 2 years of age
  Neurodevelopmental assessment using the Bayleys scale version III

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Saenz de Pipaon Marcos, Professor, Study Director — HOspital La Paz Institute for Health Research

IPD SHARING:
Plan to Share IPD: Yes
The intermediate and final data generated in the project will be uploaded to the most appropriate repositories depending on their typology and whenever possible for confidentiality issues and that does not hinder the protection of any possible intangible asset, provided that deal with Trustworthy Digital Repositories (Research Libraries Group, 2002) and follow the reference model OASIS, developed by the Consultative Committee for Space Data Systems (accredited by the ISO standard 14721:2012). In this way, these data, as well as the publications derived from the development of the project, will be deposited, among others, in the Institutional HEALTH REPository of the Carlos III Health Institute (REPISALUD, https://repisalud.isciii.es/), and in the Institutional Repository of the Ministry of Health of the Community of Madrid. Access for other researchers who may be legitimately interested will be subject in any case to their approval, complying with the requirement of open access